CLINICAL TRIAL: NCT00585455
Title: Effects of Chronic Sertraline Hydrochloride Administration on Vascular Endothelial and Autonomic Function in Patients With Chronic Heart Failure
Brief Title: Vascular Effects of Sertraline in Heart Failure
Status: Terminated | Type: Observational
Why Stopped: PI change in institution
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Stuart Katz, Yale University School of Medicine
Other Study IDs: 0410027131
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Heart Failure; Depression
Keywords: vascular endothelium; nitric oxide; depression; heart failure; vascular biology
MeSH Terms: conditions — Heart Failure; Depression | interventions — Sertraline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Chronic heart failure patients with concomitant depression
  Interventions: Drug: sertraline

INTERVENTIONS:
Drug: sertraline — open label 25-50 mg daily as tolerated

SUMMARY:
To determine the effects of chronic sertraline treatment on brachial artery flow-mediated dilation in patients with chronic heart failure and depression

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with LVEF<40%, age >21 years
* Depression requiring medical treatment with sertraline

Exclusion Criteria:

* Known intolerance of sertraline

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic heart failure patients with concomitant depression
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States